CLINICAL TRIAL: NCT07040969
Title: Spirulina-Derived Product Alleviates Oral Mucositis in Patients Undergoing Radiotherapy for Malignant Head and Neck Tumors: A Randomized Controlled Trial
Brief Title: Spirulina-Derived Product Alleviates Oral Mucositis in Patients Undergoing Radiotherapy for Malignant Head and Neck Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025(1088)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Radiation-induced Oral Mucositis
Keywords: Head & neck cancer; Radiation-induced oral mucositis; spirulina; exosome
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Spray of placebo
  Interventions: Drug: Spray of placebo; Radiation: Radiotherapy
- Experimental group (Experimental): Spray of spirulina derivatives
  Interventions: Drug: Spray of spirulina derivatives; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Spray of spirulina derivatives — An oral spray formulated with purified spirulina-derived exosomes.
  Arms: Experimental group
Drug: Spray of placebo — The placebo oral spray will be formulated with inactive ingredients matched in appearance and flavor profile to the active spirulina-derived product.
  Arms: Control group
Radiation: Radiotherapy — One of the inclusion criteria for the study was that patients with squamous carcinoma of the head and neck (including nasopharyngeal carcinoma) needed to receive either radiotherapy alone or simultaneous radiotherapy and chemotherapy.

SUMMARY:
To evaluate the efficacy and safety of Spirulina-Derived Product for prevention and treatment of oral mucositis in patients undergoing radiotherapy for malignant head and neck tumors.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of spirulina-derived product in reducing the incidence, duration, and severity of severe oral mucositis (SOM). The study primarily aims to address two questions: (1) whether spirulina-derived product can effectively prevent and mitigate radiation-induced oral mucositis, and (2) whether its use is associated with adverse events in patients undergoing radiotherapy.

Participants will be instructed to orally administer the spirulina-derived product or placebo spray four times daily, starting from the first day of radiotherapy (RT) and continuing throughout the RT course. After each spray application, patients must refrain from eating, drinking, or performing oral hygiene activities for at least 1 hour to maximize mucosal contact time of the intervention.

The study will compare the spirulina-derived product group with the placebo group to determine the potential benefits of this spirulina-based intervention in preventing and managing radiotherapy-related oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
2. Aged ≥ 18 years;
3. Eastern Cooperative Oncology Group performance status of ≤2;
4. Receiving definitive RT or postoperative adjuvant RT at a dose of 60- 72 Gy with/without concurrent chemotherapy;
5. Sign informed consent.

Exclusion Criteria:

1. Patients with known allergy to Spirulina components or severe allergic constitution;
2. Use of antibiotics, antifungal drugs, or antimicrobial mouthwash within 1 month of the study;
3. Poor oral hygiene and/or severe periodontal diseases;
4. History of head and neck radiotherapy;
5. Deemed unsuitable for the study by the investigators (concomitant with any other severe diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of severe oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks to 14.5 weeks.
  Oral mucositis is assessed by trained radiotherapists according to World Health Organization (WHO) oral toxicity Scale.The WHO Oral Toxicity Scale categorizes oral mucositis into grades 0-4, with the higher the grade the more severe the patient's oral mucositis. Grade 0 means that the oral mucosa is normal and the patient has no symptoms or signs; grade 1 means that the mucosa is erythematous with or without pain and does not interfere with eating; grade 2 means that the mucosa is erythematous and ulcerated, but still able to eat solid food; grade 3 means that the mucosa is severely ulcerated with extensive erythema and unable to eat solid food; and grade 4 means that the ulcers of the mucosa are fused together into a sheet, and their severity is so severe that it is not possible to eat.

SECONDARY OUTCOMES:
The time to onset of severe oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first day of radiotherapy to the first determination of SOM.
The duration of severe oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM.
The incidence of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale.
The time to onset of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first day of radiotherapy to the first determination of OM.
The duration of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of OM to the first instance of non-OM, without a subsequent instance of OM.
Adverse events | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version

OTHER OUTCOMES:
The longitudinal dynamics of salivary microbiota | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Unstimulated whole saliva samples will be collected via spitting method at three time points: baseline, mid-term radiotherapy (the week corresponding to 50% completion of the planned radiation fractions), and the end of radiotherapy (the final week of RT). 16S rRNA gene sequencing will be performed to assess alterations in the oral microbiota.
Taste function | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Taste strips test.
Mouth and throat soreness (MTS) scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms
Oral activities scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy. The evaluation period is approximately 6 weeks and 6.5 weeks.
  Patients report the degree to the impact of MTS on oral activities (including swallowing, drinking, eating, talking, sleeping) (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms.
Longitudinal analysis of alterations in peripheral blood immune cell profiles among patients | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Quantification of absolute counts and percentages of T cells, B cells, and NK cells in peripheral blood from patients.
Xerostomia | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Xerostomia was graded per CTCAE v5.0 (Grade 1-4), with higher grades indicating worse symptoms.
The number of patients who missed five or more consecutive radiation fractions | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  The number of patients who missed five or more consecutive radiations and the reasons for this are recorded during radiotherapy.
Analysis of inflammatory Indicators in peripheral blood | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Measurement of circulating levels of interleukin-1β (IL-1β), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) in patient peripheral blood.
Analysis of Inflammatory Indicators in Oral Saliva | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Measurement of circulating levels of interleukin-1β (IL-1β), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) in patient oral saliva.
Overall Health Status and Core Dimensions of Quality of Life | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) This instrument is a 30-item patient-reported outcome (PRO) measure designed to evaluate core aspects of health-related quality of life in cancer patients, including 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, pain, nausea and vomiting), one global health status/quality of life scale, and 6 single-item symptom measures. Scores are linearly transformed to a range of 0-100. For the functional scales and the global health status scale, higher scores indicate better functional levels or quality of life; for the symptom scales/items, higher scores indicate greater symptom burden.
Head and Neck Cancer-Specific Symptoms | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  The EORTC QLQ-H&N35 is a patient-reported outcome (PRO) instrument specifically designed to assess disease-related symptoms and treatment-related side effects in patients with head and neck cancer. It comprises 35 items, organized into seven multi-item subscales (pain, swallowing, senses, speech, social eating, social contact, and sexuality) and eleven single-item measures (such as dental problems, problems opening mouth, sticky saliva, coughing, etc.). All subscale and single-item scores are linearly transformed to a 0-100 scale using a standardized scoring algorithm. Interpretation of Scores: For all subscales and single items, higher scores represent more severe symptoms or greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No